CLINICAL TRIAL: NCT07405242
Title: A Single-arm, Open-label, Multicenter Clinical Study Evaluating the Safety and Efficacy of Endovascular Treatment for Retrograde Dissections Involving the Ascending Aorta That Are Not Suitable for Open Surgery. （RADIAL)
Brief Title: Retrograde Ascending Dissection: Intraluminal Aortic Therapy
Acronym: RADIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RX-2025-004
Record Dates: First submitted 2026-01-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Ascending Aortic Dissection
MeSH Terms: conditions — Dissection, Ascending Aorta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular treatment of aortic dissection (stent implantation) (Experimental)
  Interventions: Device: Endovascular treatment of aortic dissection (stent implantation)

INTERVENTIONS:
Device: Endovascular treatment of aortic dissection (stent implantation) — Endovascular treatment of aortic dissection (stent implantation)

SUMMARY:
This study is a single-arm, open-label, multi-center clinical trial evaluating the safety and efficacy of endovascular treatment for retrograde dissection involving the ascending aorta that is not suitable for open surgery. The aim is to assess the short-term (30 days) and medium- to long-term (6 months and 12 months) safety and efficacy of endovascular treatment in patients with retrograde dissection involving the ascending aorta who are not suitable for open surgery. The study plans to include patients with dissection confirmed by imaging, with the tear located in the aortic arch or descending aorta and extending retrogradely to the ascending aorta, and the most distal segment of the dissection is at least 2 cm away from the coronary artery ostia. These patients have been evaluated by cardiac surgery and found to be unsuitable for open surgery, with significant risks or risks outweighing benefits associated with open surgery. This is a single-arm, open-label, multi-center study, and no blinding or randomization will be used, nor will stratification factors be set. After successful screening, the subjects will undergo endovascular treatment for aortic dissection (stent implantation) during the operation. The subjects will be followed up for one year after the operation, and the safety and efficacy of endovascular treatment for retrograde dissection involving the ascending aorta will be evaluated based on the subjects' survival status, the occurrence of surgery and disease-related complications, and the recovery of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the clinical trial; The individual fully understands and is informed of this study and has signed the informed consent form; Willing to follow and be able to complete all trial procedures
* Age ≥ 65 years old, both male and female are eligible
* Confirmed by imaging to be retrograde tear aortic dissection, that is, the tear site is located at the aortic arch or descending aorta, and the retrograde tear involves the ascending aorta. The farthest segment of the dissection tear is ≥ 2 cm from the coronary artery outlet
* Evaluation by cardiac surgery indicates that open surgical treatment is not suitable, performing open surgery poses significant risks or the risks outweigh the benefits
* Arterial access conditions are permitted, without severe stenosis or distortion, and the stent delivery system can be smoothly introduced;

Exclusion Criteria:

* Severe organ ischemia or functional failure, which, after assessment, is considered to have an extremely poor prognosis and cannot benefit from endovascular treatment, such as extensive cerebral infarction or cerebral hemorrhage, resulting in irreversible severe neurological deficits, acute extensive ischemic necrosis of the mesenteric arteries, acute liver and kidney failure;
* Planned to undergo aortic valve repair/replacement or coronary artery interventional therapy within 30 days;
* Mechanical heart valve present at the aortic valve position;
* Aortic valve regurgitation degree ≥ 3+ or 4+;
* Known severe allergy to contrast agents or stent materials (such as nickel-titanium alloys, polyester, etc.);
* Severe systemic infection that may lead to infection after stent implantation;
* Severe coagulation dysfunction, which, after correction, still cannot meet the surgical requirements, or has bleeding tendencies;
* Complicated with other serious diseases or malignant tumors, with a predicted survival period of less than 12 months;
* Pregnant or lactating women;
* With mental illness or cognitive impairment, unable to understand and cooperate with the study;
* Already participating in other ongoing interventional clinical studies;
* Other situations judged by the investigator as not suitable for inclusion in the study;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The death events and major adverse cardiovascular and cerebrovascular events (MACCE) caused by any reason within 30 days after endovascular treatment, as well as their incidence rates | 30 days

SECONDARY OUTCOMES:
The incidence rate of surgery-related complications | 12 months
Success rate of one-year stent implantation technique | 12 months
The all-cause mortality rates for 6 months and 12 months | 12 months
The incidence rates of major adverse cardiovascular and cerebrovascular events within 6 months and 12 months | 12 months
The rates of re-intervention for aortic dissection within 6 months and 12 months | 12 months
The incidence rates of complications related to aortic dissection for 6 months and 12 months | 12 months
Aortic imaging remodeling assessment: Changes in the true lumen diameters of the ascending aorta, aortic arch, and descending aorta at 6 months and 12 months after surgery, and the proportion of false lumen reduction or complete thrombosis | 12 months
Quality of life assessment: The SF-36 scale was used to evaluate the patients' quality of life scores before the surgery, 6 months after the surgery, and 12 months after the surgery. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University Medical School Affiliated Ruijing Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF